CLINICAL TRIAL: NCT00165594
Title: Non-Randomized, Open, Uncontrolled, Dose Comparison Study of E7070 in Patients With Gastric Cancer
Brief Title: A Study of E7070 in Patients With Gastric Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was completed.
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7070-J081-217
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; Phase I; Phase IIa; E7070; Indisulam; Pharmacogenomic; 2C19
MeSH Terms: conditions — Stomach Neoplasms | interventions — N-(3-chloro-7-indolyl)-1,4-benzenedisulphonamide

INTERVENTIONS:
Drug: E7070

SUMMARY:
Phase I study:

To investigate primary objective (maximal tolerated dose and dose-limiting toxicity) and secondary objectives (pharmacokinetics, safety, estimation of a recommended dose, and anti-tumor effect by evaluable case) of E7070 in patients with gastric cancer who are extensive or intermediate metabolizer type (EM/IM) to CYP2C9 and CYP2C9 by intravenously administering once every 3 weeks.

Phase IIa study:

To investigate primary objective (response rate for efficacy assessment) and secondary objectives (frequency and severity of adverse drug reactions, and pharmacokinetics) of E7070 in patient with gastric cancer who are EM/IM type by intravenously administering once every 3 weeks.

ELIGIBILITY:
Inclusion Criteria (Phase I):

* Patients who are histologically or cytologically confirmed to have gastric cancer.
* Patients who are non-responder to existing treatments with proved efficacy for gastric cancer, but any further effect is no longer expected with existing treatments.
* Patients who are aged ≥20 years and <75 years at the time of registration.
* Patients graded as 0 - 2 of the Eastern Cooperative Oncology Group (ECOG) Performance status (PS)
* Patients who can be hospitalized between the beginning of the study treatment and the end of the first cycle.
* Patients with well-maintained functions of major organs (bone marrow, liver, kidney, and lung).

  1. WBCl count: ≥3,000/mm3, ≤12,000/mm3
  2. Neutrophil count: ≥2,000/mm3
  3. Platelet count: ≥100,000/mm3
  4. Hemoglobin: ≥9.0 g/dL
  5. Aspartate aminotransferase (AST): ≤2.5 times the upper limit of normal range at the study site
  6. Alanine aminotransferase (ALT): ≤2.5 times the upper limit of normal range at the study site
  7. Total bilirubin: ≤1.5 times the upper limit of normal rage at the study site
  8. Serum creatinine: ≤1.5 times the upper limit of normal range at the study site
  9. Partial pressure oxygen in arterial blood: ≥65 torr
* Patients who are EM/IM regarding CYP2C9 and CYP2C19
* Patients who consented to participate in this study with a written consent form
* Patients who have no carry-over adverse drug reaction(s) that affect the evaluation of previous treatments and safety of E7070 after the completion of the previous treatment. Required periods of wash-out from the end of previous treatment to the beginning of the study treatment are as follows:

  1. Chemotherapy, endocrinotherapy, immunotherapy, radiotherapy, surgical therapy, and other investigational products: 4 weeks
  2. Nitrosourea agents and mitomycin C: 6 weeks
  3. Blood transfusion, blood preparations, and hematopoietic preparations including G-CSF preparation: 2 weeks
* Patients who are expected to survive for at least 3 months from the beginning of the study treatment.

Exclusion Criteria (Phase I):

* Patients with systemic infectious disease.
* Patients with a large volume of pleural effusion, ascites, or pericardial effusion that requires drainage.
* Patients who have brain metastasis with clinical symptoms.
* Patients who have a clinically significant mental disorder, attack, or central nervous-related disorder.
* Patients who meet any of the following serious complications:

  1. Ischemic heart disorders or heart diseases including arrhythmia that requires medical treatment (excluding left ventricular hypertrophy, mild left ventricular load, or mild right bundle branch block accompanied with hypertension).
  2. Myocardial infarction within 6 months.
  3. Hepatic cirrhosis.
  4. Interstitial pneumonia or pulmonary fibrosis.
  5. Gastrointestinal fresh hemorrhage that requires repeated blood transfusion.
  6. Uncontrolled diabetes mellitus (hemoglobin Alc (HBAlc): ≥8.0 %)
* Patients whose NYHA classification is II - IV.
* Patients who meet any of the following items regarding prolonged QT/QTc intervals:

  1. A history of prolonged QT/QTc intervals (male: QTc > 450 ms, female: QTc > 470 ms (Bazett's correction))
  2. At the time of registration: QTc > 500 ms (Bazett's correction)
  3. A history of serious arrhythmia including Torsades de pointes
* Patients who require nutrition support using intravenous hyper alimentation (IVH) or enteral nutrition.
* Patients who have a history of hypersensitivity to sulfonamide.
* Premenopausal women who are currently pregnant, breastfeeding, or childbearing potential. Premenopausal women of childbearing potential are defined as women with less than a 12-month elapse after the last menstruation, and their pregnant test is positive or not performed at the time of registration, or they do not consent for using an appropriate contraceptive method.
* Male patients who have no intention of contraception.
* Patients on a coumarin agent or who has taken it within 2 weeks before starting the study treatment.
* Patients who are currently taking an agent that is known to cause prolonged QT/QTc intervals.
* Patients who are positive for a test of human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus surface antigen (HBs antigen).
* Patients who have a history of drug or alcohol abuse.
* Patients who continuously require systemic treatment with a steroid during the study period.
* Patients who are presently participating in another clinical study.
* Patients who are judged to be ineligible for participating in this study by the investigator or sub investigator.

Inclusion Criteria (Phase IIa):

* Patients who are histologically or cytologically proved efficacy for gastric cancer.
* Patients unable to undergo resection or with recurrence of cancer.
* Patients with evaluable lesions based on RECIST.
* Patients treated with 1 or 2 regimens of previous chemotherapy for gastric cancer (at least 1 regimen using fluorouracil agent). Adjuvant chemotherapy with an oral pyrimidine fluoride agent is not included in the number of previous regimen.
* Patients who are aged ≥20 years and <70 years.
* Patients graded as 0 - 2 as the Eastern Cooperative Oncology Group (ECOG) Performance status (PS)
* Patients who can be hospitalized from the beginning of study treatment to the end of the first cycle.
* Patients with well-maintained functions of major organs (bone marrow, liver, kidney, and lung).

  1. WBC count: ≥3,000/mm3, ≤12,000/mm3
  2. Neutrophil count: ≥ 2,000/mm3
  3. Platelet count: ≥100,000/mm3
  4. Hemoglobin: ≥9.0 g/dL
  5. Aspartate aminotransferase [AST]: ≤2.5 times the upper limit of normal at the center
  6. Alanine aminotransferase [ALT]: ≤2.5 times the upper limit of normal at the center
  7. Total bilirubin: ≤1.5 times the upper limit of normal at the center
  8. Serum creatinine: ≤1.5 times the upper limit of normal at the center
  9. Partial pressure oxygen in arterial blood: ≥65 torr
* Patients who are EM/IM regarding CYP2C9 and CYP2C19
* Patients who consented to participate in this study with a written consent form.
* Patients who have no carry-over adverse drug reaction(s) that affect the evaluation of previous treatment and safety of E7070 after the completion of the previous treatment. Required periods of wash-out from the end of previous treatment to the beginning of study treatment are as follows.

  1. Chemotherapy, endocrinotherapy, immunotherapy, radiotherapy, surgical therapy, and other investigational products: ≥4 weeks
  2. Nitrosourea agents and mitomycin C: ≥6 weeks
  3. Blood transfusion, blood preparations, and hematopoietic preparations including G-CSF preparation: ≥2 weeks
* Patients who are expected to survive for at least 3 months from the beginning of treatment with the investigational product.

Exclusion Criteria (Phase IIa):

* Patients with systemic infectious disease.
* Patients with severe peritoneal dissemination that meet any of the following items.

  1. Clinical sign of ileus or sub ileus
  2. Worse than moderate ascites (beyond over pelvic cavity)
  3. Clear peritoneal dissemination confirmed with enema
* Patients with a large volume of pleural effusion, ascites, or pericardial effusion that require drainage.
* Patients who have brain metastasis with clinical symptoms
* Patients who have clinically significant metal disorder, attack, or central nervous-related disorder.
* Patients who meet any of the following serious complications:

  1. Ischemic heart disease or other heart disease including arrhythmia that require medical treatment (excluding left ventricular hypertrophy, mild left ventricular load, or mild right bundle branch block accompanied with hypertension)
  2. Myocardial infarction within 6 months
  3. Hepatic cirrhosis
  4. Interstitial pneumonia or pulmonary fibrosis
  5. Gastrointestinal fresh hemorrhage that requires repeated blood transfusion
  6. Uncontrolled diabetes mellitus (hemoglobin Alc (HbAlc) ≥ 8.0 %)
* Patients whose NYHA classification is II - IV.
* Patients who meet any of the following items regarding prolonged QT/QTc intervals.

  1. A history of prolonged QT/QTc intervals (male: QTc > 450 ms, female: QTc > 470 ms (Bazett's correction))
  2. At the time of registration: QTc > 500 ms (Bazett's correction)
  3. A history of serious arrhythmia including Torsades de pointes
* Patients who require nutrition support with intravenous hyper alimentation (IVH) or enteral nutrition.
* Patients who have a history of hypersensitivity to sulfonamide.
* Patients with active multiple malignant tumor (including disease-free interval within 5 years)
* Premenopausal women of currently pregnant, breastfeeding or childbearing potential. Premenopausal women of childbearing potential are defined as women with less than a 12-month elapse after the last menstruation and pregnant test is positive or not performed at the time of registration, or they do not consent for an appropriate contraceptive method.
* Male patients who have no intention of doing contraception.
* Patients who are currently taking a coumarin agent or has taken it within 2 weeks before the beginning of study treatment.
* Patients who are currently taking an agent that is known to cause prolonged QT/QTc intervals.
* Patients who are positive for a test of human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus surface antigen (HBs antigen).
* Patients who have a history of drug or alcohol abuse
* Patients who continuously require systemic treatment with a steroid during the study period.
* Patients who are presently participating in another clinical study.
* Patients who are judged to be ineligible for participating in this clinical study by the investigator or sub investigator

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-02; Primary Completion 2006-07 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Phase I study:
Dose-limiting toxicity (DLT)
Phase IIa study:
Response rate based on Response Evaluation Criteria in Solid Tumors (RECIST)

SECONDARY OUTCOMES:
Phase I study:
Plasma E7070 concentration.
Adverse event, adverse drug reaction, laboratory parameter, and vital sign.
Anti-tumor effect based on (RECIST).
Phase IIa study:
Adverse drug reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuo Watanabe, Study Director — Eisai Co., Ltd - Development Clinical Research Department. Clinical Research Center
Locations (5):
- Japan (5):
  - Kashiwa, Chiba
  - Sagamihara-shi, Kanagawa
  - Takatsuki-shi, Osaka
  - Sunto-gun, Shizuoka
  - Chuo-ku, Tokyo